CLINICAL TRIAL: NCT04619212
Title: A Pre-market, Prospective, Comparative, Concept Proofing, Study Evaluating if Mothers Who Are Both Breastfeeding and Pumping in the First Days After Delivery Report Improved Comfort Levels With the New Symphony Program Card INITIATE 2.0 Program Compared With the Current Standard of Care, the Symphony Plus Program Card.
Brief Title: Initiate Study Evaluating if Mothers Who Are Both Breastfeeding and Pumping in the First Days After Delivery Report Improved Comfort Levels With the New Symphony Program Card
Acronym: Initiate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medela AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MHM_2003
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2021-09

CONDITIONS: Breast Pumping
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: 2 different groups, where 1 group does SoC (comparator device), the second uses the new device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): Standard of Care
  Interventions: Device: breast pumping as per SoC but on new software for the pump
- new device (Other): new device
  Interventions: Device: breast pumping as per SoC but on new software for the pump

INTERVENTIONS:
Device: breast pumping as per SoC but on new software for the pump — breast pumping as per SoC but on new software for the pump

SUMMARY:
The study hypothesizes that mothers who are both breastfeeding and pumping in the first days report improved comfort levels with the new Symphony program card INITIATE 2.0 compared to the standard of care.

DETAILED DESCRIPTION:
This study aims to investigate whether the proposed changes to the INITIATE 2.0 program card lead to an improvement in comfort during pumping as well as increased milk removal during a pumping session. The results of this study will provide important information that a) validates the proposed changes as well as b) builds clear recommendations for which vacuum level should be used for Symphony program cards in this population.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 18 years old
* Infant was born maximum 4 (96 hours) days ago
* Subject aims to provide breastmilk for the baby through breastfeeding.
* At least 50% of the milk removal sessions in the last 24hrs were breastfeeds.
* Subject has an indication to pump for reasons
* The subject signs the informed consent documentation

Exclusion Criteria:

* Woman is exclusively pumping
* Woman is experiencing a mastitis event
* Woman is still breastfeeding with the previous child
* Woman has been breastfeeding in the last 6 months
* Woman received morphine pain medication in the last 8 hours

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women can produce human milk
Enrollment: 80 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | during the 20 minutes pumping procedure. this is the only visit and task for the patient.
  Number of patients with adverse events & description
Comfort while pumping | Within the 20 minutes pumping procedure. this is the only visit and task for the patient.
  Assessed by the necessity of reducing the vacuum strength during pumping (binary outcome). It is expected that mothers should not need to change the vacuum strength when using the new program card

SECONDARY OUTCOMES:
Performance of the new software | during the 20 minutes pumping procedure. this is the only visit and task for the patient.
  The output milk volume will be measured between the standard of care (pumping) approach and the new program card INITIATE 2.0

CONTACTS AND LOCATIONS:
Overall Officials: Fedde Scheele, Principal Investigator — Study team
Locations (1):
- OLVG Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
individual data is not shared.

REFERENCES:
- [Derived] Nicole Manshanden TM, Prime DK, Scheele F, Velzel J. Impact of a Modified Breast Pump Suction Pattern on Milk Yield During the Initiation of Lactation: A pilot study. J Perinat Neonatal Nurs. 2025 Nov 24. doi: 10.1097/JPN.0000000000000975. Online ahead of print. PMID 41276904
- [Derived] Manshanden TMN, Prime DK, Scheele F, Velzel J. An evaluation of patient comfort levels during expression with a modified pumping program: a prospective proof of concept study. Front Glob Womens Health. 2024 Apr 19;5:1378263. doi: 10.3389/fgwh.2024.1378263. eCollection 2024. PMID 38707635